CLINICAL TRIAL: NCT01623973
Title: Impact of the Restriction of the Non Paretic Upper Limb in Rehabilitation of Patients Post-stroke:Randomized Clinical Trial
Brief Title: Impact of Restriction of the Non Paretic Upper Limb Rehabilitation of Patients a With Stroke:Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Luciana B. dos Santos, PT, Impact of restriction of the non-paretic upper limb rehabilitation of patients after stroke: a randomized blinded clinical trial, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-2012-MDTR, Brazil
Record Dates: First submitted 2012-06-12; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Stroke
Keywords: hemiparetic; cognitive; balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With restraint (Experimental): The group with restraint underwent specific training of paretic upper limb and use of restraint.
  Interventions: Other: specific training of paretic upper limb
- no restraint (Active Comparator): The group control "without restraint" submitted only to the specific training of paretic upper limb
  Interventions: Other: specific training of paretic upper limb

INTERVENTIONS:
Other: specific training of paretic upper limb — nineteen individuals with chronic stroke was randomly assigned, after the first evaluation, into two groups: group without restriction (G1), subject only to the specific training of paretic UL, and restricted group (G2), which underwent specific training of paretic UL and use of the restriction of non paretic UL. The volunteers were evaluated before the beginning of the interventions, and the next day after completion of the 12 therapy sessions through the Fugl-Meyer Assessment

SUMMARY:
To evaluate whether the restriction of the non paretic upper limb (UL) is a factor that could interfere at the sensorimotor UL recovery for chronic stroke subjects and to verify the impact on daily function, quality of life. In this pilot, randomized, blind and allocation concealment clinical trial, nineteen individuals with chronic stroke was randomly assigned, after the first evaluation, into two groups: group without restriction (G1), subject only to the specific training of paretic UL, and restricted group (G2), which underwent specific training of paretic UL and use of the restriction of non paretic UL

ELIGIBILITY:
Inclusion Criteria:

* ability to actively extend at least 10° at the metacarpophalangeal the wrist;
* more than 6 months post onset of stroke;

Exclusion Criteria:

* Mini-Mental State Examination;
* no excessive spasticity in any joints of the affected.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To investigate the impact that the restriction of non-paretic upper limb recovery would have on sensorimotor with Fugl-Meyer Scale | 1 year
  Upper extremity motor impairment was evaluated using the Fugl-Meyer Assessment Scale (FM).This scale has a total score of 66 points for upper limbs, reflecting a mild motor impairment (≥ 50), moderate to severe (50-20) and severe (< 20).

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | 1 year
  The FIM consists of 18 items divided into 6 subscales measuring self-care, sphincter control, transfer, locomotion, communication, and social cognition ability. Each item is rated from 1 to 7 based on the required level of assistance to perform the basic ADL (maximum score, 126). Higher scores demonstrate greater independent participation in daily activities.